CLINICAL TRIAL: NCT05242068
Title: Can Veinlite Reduce Complications of Peripheral Intravenous Catheter Placement in Children: Preliminary Results.
Brief Title: Can Veinlite Reduce Complications of Peripheral Intravenous Catheter Placement in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ayşe Kahraman, associate professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E.314064
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Catheterization; Pain; Complication
Keywords: pain; children; vein imaging device; intravenous complications
MeSH Terms: conditions — Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study was a prospective randomized controlled clinical study of children treated in a pediatric surgical ward who required PIC. The aim of the research was to evaluate whether the Veinlite would prevent catheter-related complications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care of group (Other): Patients in standard care of group received traditional peripheral intravenous catheterization
  Interventions: Other: Standard care
- Veinlite group (Experimental): Patients in veinlite group received peripheral intravenous catheterization with Veinlite
  Interventions: Device: Veinlite

INTERVENTIONS:
Device: Veinlite — Use of vein imaging device for visualization of veins during peripheral IV placement
  Arms: Veinlite group
Other: Standard care — Patients received standard intravenous catheterization.
  Arms: Standard care of group

SUMMARY:
This study was conducted to investigate the use of Veinlite LED+ (TransLite, Sugar Land, Tex) to assist with PIC placement. The Veinlite uses LED (light-emitting diode) lights to enhance the visualization of veins by using orange and red color that are absorbed in venous blood.

The investigators' hypothesis for this study was that the vein imaging would reduce the complications related to catheter and the pain that the participants would feel.

DETAILED DESCRIPTION:
Peripheral Intravenous Catheterization (PIC) introduces multiple risks and potential morbidities. Patients with PIC-associated complications have longer length of stay, higher clinical and economic burden, and greater risk of death than patients without. The most serious complications due to intravenous (IV) catheters are infiltration and extravasation.

The primary endpoint was to evaluate whether Veinlite LED+ would prevent catheter-related complications.

The secondary endpoint were;

1. to evaluate the efficacy of the vein imaging device on pediatric pain during intravenous catheterization
2. to evaluate the efficacy of the vein imaging device on catheter dwell time.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 5 and 18
* Children with DIVA (Difficult intravenous access score) score 4 or more
* That the child and the parent speak Turkish

Exclusion Criteria:

* needing urgent treatment
* a critical health condition
* That the child or the parent has a communication problem

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Children in both the Standard care of group and Veinlite group were to be stratified into three age groups: 5 to 9, 10 to 14 and 15 to 18
Enrollment: 139 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
Reducing number of complications related with peripheral intravenous catheter | Duration of catheter dwell time (up to 168 hours)
  Reducing number of complications related with peripheral intravenous catheter during treatment

SECONDARY OUTCOMES:
Pain scores during peripheral intravenous catheterization | Immediately after IV placement
  Pain scores by child, nurse, and parent. In this study, numerical rating score was used for determine pain level. The numeric rating scale is one of the most commonly used to obtain self-reports of pain intensity in school-age children, adolescents, and adults. The numerical rating scale (NRS) requires the child to rate her/his pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Catheter dwell time | Up to 168 hours (1 week)
  Intravenous catheter survival time during the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No